CLINICAL TRIAL: NCT00496171
Title: A Phase I Hexaminolevulinate (HAL) Dose-Finding Study Applying Different Formulations to the Cervix in Healthy Volunteers
Brief Title: Phase I Study of HAL Formulations Applied to the Cervix in Healthy Volunteers
Status: Terminated | Type: Observational
Sponsor: Photocure (Industry)
Other Study IDs: PC CE102/07
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2009-01-16 (Estimated); Status verified 2009-01

CONDITIONS: Healthy

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of the study is to determine the most effective formulation of HAL for release of hexaminolevulinate to the cervical epithelium at different doses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, pre-menopausal female volunteers

Exclusion Criteria:

* Acute or chronic disease which could influence the study results

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Claes G Tropé, MD PhD, Principal Investigator — Riks-Radium University Hospital
Locations (1):
- Riks-Radium University Hospital, Oslo, Norway